CLINICAL TRIAL: NCT04745208
Title: The Effect of Simulation-Based Training on the Preparedness and Burden of Caregiver of Patients With Burns: A Randomised Controlled Study
Brief Title: Simulation-Based Training on the Preparedness and Burden of Caregiver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Sabri Karahan, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KA-19021
Record Dates: First submitted 2020-08-12; First posted 2021-02-09 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Burns
Keywords: burn; simulation; burden of care; readiness for caregiving.; caregiver
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: Simulation-based education will be performed after the standard discharge training with the intervention group. The control group will receive only the standard discharge education
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be masked in the clinical trial. One of the investigators will enter the data by giving "a" for control group and "b" for intervention group. So that, the outcome assessor will not have knowledge which group is exposed to intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard discharge education (No Intervention): The control group will receive only the standard discharge education.
- standard discharge education+Simulation based education (Experimental): The intervention group will receive standard discharge education and then simulation based education will be performed
  Interventions: Behavioral: Simulation based education

INTERVENTIONS:
Behavioral: Simulation based education — high fidelity simulation with moulage
  Arms: standard discharge education+Simulation based education

SUMMARY:
Major burn injuries are serious traumas that cause physical and psychological problems. The acute period that begins with admission to the hospital is followed by a rehabilitation period that lasts for months or even years. The main goal in the acute care of the patient in hospital is to discharge the patient from the hospital as soon as possible, with the least morbidity, functional and cosmetic loss. The care of the patient in rehabilitation period continues at home, and the home care is provided by informal caregivers. Due to the physiological and psychological changes occurring in the patient with burns, the informal caregiver has important duties such as; helping with or doing feeding, wound care, personal care, organizing household chores, providing economic, medical and psychological support. So that, informal caregivers may experience lack of information and anxiety. Nurses should include the informal caregivers in discharge education to meet the information requirement of them, to prepare them for home care and to reduce anxiety of home care. The basis of discharge education is to help individual to cope with the problems related to the disease and to maintain individual care. Nurses, who play a key role in discharge education, have been keeping up with the change over the years and trying to maintain the effectiveness of education by various methods. The educational environment enriched with different technological tools and materials used in the field of education makes it easier to provide a change of behavior in the desired direction in the learner. A controlled and safe simulation environment ensures patient safety at all times, while ensuring that training is tailored specifically to the needs of the trained. Simulation gives caregivers an opportunity to manage stressful medical events in a risk-free environment, which allows healthcare providers to be involved in and manage the family's traditional education when it comes to caring and teaching families. When the literature on increasing the preparedness of the caregivers for care, and thus reducing the burden of care, no studies evaluating the simulation-based training for informal caregivers were found. This study was needed with the idea that simulation-based training, which is provided with a high fidelity of moulage, will help the caregiver to understand the burn care easily, to be ready for care and therefore to reduce the burden of care.

DETAILED DESCRIPTION:
Method:

The study was designed as a randomised controlled study with the control group in order to determine the effect of simulation-based training applied to the caregivers of burn patients on their preparedness for care and caregiving burden. The research will be conducted in the Burn Unit of Hacettepe University Adult Hospital and Burn Center of Gulhane Training and Research Hospital. The population of the research includes caregivers of adult patients admitted to Hacettepe University Adult Hospital Burn Unit and Burn Center of Gulhane Training and Research Hospital after 02.02.2021 and have treatment in inpatient or outpatient clinics. Since there is no similar research in the literature, sample size was not calculated. At the end of the study, power analysis will be done to evaluate the adequacy of the sample size. In the study, participants in the intervention group and control group will be assigned by block randomization method and each block will consist of 4 caregivers and 6 blocks will be formed. The data sheets of the research are Caregivers Information Form, Preparedness for Caregiving Scale, Caregiving Burden Scale and Post-Discharge Assessment Form for Burn patients. In addition, the Questionnaire for the Burn patients will be used to obtain information about the burn patients.

Implementation of study:

The control group will receive only the standard discharge education. Simulation based education will be performed after the standard discharge training with the intervention group. The preparedness of caregivers before and after both training will be assessed. The burden of caregiving will be assessed during the first and third months of care.

Collection of Data:

In order to test the understandability of standard discharge training, training will be provided to 3 patient relatives. The presentation of the training will be organized according to the feedback received.

After the pre-application of the simulation scenario in the laboratory environment 3 times, the necessary changes will be made on the scenario and the final version will be given.

Data collection tools will be applied on the both group, unrecognized questions and corrections will be made on missing items. Individuals participating in these preliminary studies will not be included in the study.

Percentage, mean, standard deviation will be used in the evaluation of the data. Chi-square, Fisher's exact test, independent paired T-test and Mann-Whitney U test will be used for comparison between groups and within groups. p <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Caring for patients with burn during the study
* Being over 18 years old
* Agree to participate voluntarily in the study
* To communicate
* Not having a diagnosed mental problem
* The burn patient he/she cares for is over the age of 18, inpatient treatment in the burn unit, no communication problem, no diagnosed mental problem, no additional problem (fracture, paralysis, etc.) except burn.
* At least 5 days to be discharged from the burns patient,
* Not being a healthcare professional
* Not caring for another family member, except burn patients.

Exclusion Criteria:

* Loss of life of the burned individual and/or caregiver during the study.
* The participant declares that he/she wants to leave at any stage of the study.
* Not participating in data collection in the first and third months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-13 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
caregiving burden | from first month until third month
  The caregiver burden score will be assessed by Burden Scale for Family Caregivers.
Preparedness of care | First assessment at time of acceptance of the study -2 day after education
  The readiness of caregiving will be assessed at the time of acceptence and post-training education by Preparedness for Caregiving Scale.

SECONDARY OUTCOMES:
Burn Patient Fallow Up | 3 months
  Burn patients will be fallowed from through 3 months and complications, rehospitalizations number, etc. will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Zahide Tuncbilek, Asst. Prof., Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cook DA, Hatala R, Brydges R, Zendejas B, Szostek JH, Wang AT, Erwin PJ, Hamstra SJ. Technology-enhanced simulation for health professions education: a systematic review and meta-analysis. JAMA. 2011 Sep 7;306(9):978-88. doi: 10.1001/jama.2011.1234. PMID 21900138
- [Background] Deshpande, O. N., Puri, V., Vora, S. S., Shende, N. N., & Choudhary, S. C. (2012). Socio-economic burden of burns: How do the families of patients cope? Indian journal of burns, 20(1), 48.
- [Background] Evgeniou E, Loizou P. Simulation-based surgical education. ANZ J Surg. 2013 Sep;83(9):619-23. doi: 10.1111/j.1445-2197.2012.06315.x. Epub 2012 Oct 22. PMID 23088646
- [Background] Faydali, S., & Bayraktar, N. (2011). Yanıklı Hastaların ve Yakınlarının Taburculuk Sonrası Bilgi Düzeylerinin Belirlenmesi. Turkish Journal of Research & Development in Nursing, 13(1).
- [Background] Fletcher JD, Wind AP. Cost considerations in using simulations for medical training. Mil Med. 2013 Oct;178(10 Suppl):37-46. doi: 10.7205/MILMED-D-13-00258. PMID 24084304
- [Background] Grasel, E., Chiu, T., & Oliver, R. (2003). Development and validation of the Burden Scale for Family Caregivers. Toronto: Comprehensive Rehabilitation and Mental Health Services.
- [Background] Jutten LH, Mark RE, Maria Janssen BWJ, Rietsema J, Droes RM, Sitskoorn MM. Testing the effectivity of the mixed virtual reality training Into D'mentia for informal caregivers of people with dementia: protocol for a longitudinal, quasi-experimental study. BMJ Open. 2017 Aug 21;7(8):e015702. doi: 10.1136/bmjopen-2016-015702. PMID 28827242
- [Background] Sullivan-Bolyai S, Bova C, Lee M, Johnson K. Development and pilot testing of a parent education intervention for type 1 diabetes: parent education through simulation-diabetes. Diabetes Educ. 2012 Jan-Feb;38(1):50-7. doi: 10.1177/0145721711432457. Epub 2012 Jan 5. PMID 22222512
- [Background] Tofil NM, Rutledge C, Zinkan JL, Youngblood AQ, Stone J, Peterson DT, Slayton D, Makris C, Magruder T, White ML. Ventilator caregiver education through the use of high-fidelity pediatric simulators: a pilot study. Clin Pediatr (Phila). 2013 Nov;52(11):1038-43. doi: 10.1177/0009922813505901. PMID 24137039
- [Background] Ulusoy N, Graessel E. Subjective burden of family caregivers with Turkish immigration background in Germany : Validation of the Turkish version of the Burden Scale for Family Caregivers. Z Gerontol Geriatr. 2017 Jun;50(4):339-346. doi: 10.1007/s00391-016-1044-y. Epub 2016 Jun 21. PMID 27323761
- [Background] Zwicker, D. (2010). Try this: best practices in nursing care to older adults. Preparedness for caregiving scale. Hartford Institute for Geriatric Nursing, New York University of Nursing. Retrieved January, 15, 2011.